CLINICAL TRIAL: NCT02000895
Title: Early Detection of Progressive Kidney Disease in Preterm Infants
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: The Gerber Foundation (Other); Micah Batchelor Foundation (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Marissa DeFreitas, Associate Professor of Pediatrics, University of Miami
Other Study IDs: 20100986; 66787R (Other Grant/Funding Number: Gerber Foundation); 701170 (Other Grant/Funding Number: Micah Batchelor Foundation); 5KL2TR002737-04 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-12-04 (Estimated); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Urine Cord Blood Umbilical cords
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infants born preterm and of low birth weight are known to be at increased risk for early onset of cardiovascular and renal disease in adult life. This has been related to low nephron mass due to inadequate or early termination of glomerulogenesis in utero and during the perinatal period. Risks for subsequent development of hypertension and kidney disease include proteinuria, excessive weight gain during early life with insulin resistance and supplemental high calorie feedings. The long-term goal is for early diagnosis of those infants who are at risk for future development of hypertension and kidney disease so that the investigators might intervene to potentially avert progression to adult disease. The objective of this clinical trial is to acquire data on the natural history of neonatal kidney function and size in infants born preterm during the first 2 years of life. This will be done through the use of standard serum and urine markers as well as non-invasive ultrasound technology. The central hypothesis of this clinical trial is that a subgroup of patients born preterm and of low birth weight will demonstrate early markers of kidney injury including elevated serum cystatin C, proteinuria and low kidney size. This hypothesis has been formulated on the basis of preliminary data from our group studying this question retrospectively in older children born prematurely who have developed overt kidney disease. The rationale for the proposed research is to develop early serum and demographic markers of pre-clinical kidney disease so that early intervention can occur. The proposed clinical trial is innovative because it will investigate the risk factors for kidney dysfunction at a pre-clinical stage with the idea of gaining more knowledge regarding therapeutic interventions. In addition, the study will assess serum cystatin C as a surrogate test for glomerular filtration rate which could indicate worsening kidney function at an earlier stage than serum creatinine.

The proposed research is significant because it is expected to identify at-risk patients for future renal impairment and to prospectively monitor the persistence of proteinuria and its effect on kidney function in the short term.

DETAILED DESCRIPTION:
Objectives and Hypotheses:

Infants born preterm and of low birth weight are known to be at increased risk for early onset of cardiovascular and renal disease in later life. This has been related to low nephron mass due to inadequate or early termination of glomerulogenesis in utero and during the perinatal period. Risks for subsequent development of hypertension and kidney disease include excessive weight gain during early life with insulin resistance and supplemental high calorie feedings.

Specific Aims The long-term goal is for early diagnosis of those infants who are at risk for future development of hypertension and kidney disease so that investigators might intervene to potentially avert progression to adult disease. The objective of this clinical trial is to acquire data on the natural history of neonatal kidney function and size in infants born preterm during the first year of life. This will be done through the use of standard serum and urine markers as well as non-invasive ultrasound technology. The central hypothesis of this clinical trial is that a subgroup of patients born preterm will demonstrate early markers of kidney injury including elevated serum cystatin C, proteinuria and hypertension. This hypothesis has been formulated on the basis of preliminary data from the group studying this question retrospectively in older children born prematurely who have developed overt kidney disease. The rationale for the proposed research is to develop early serum and demographic markers of pre-clinical kidney disease so that early intervention may occur.

Study Design. This is a single-center case-controlled prospective observational study with the rationale of evaluating parameters of renal function including proteinuria, microalbuminuria and cystatin C in preterm infants and associating this with kidney size and blood pressure during the first 10 years of life. Demographics including race, gender and growth will provide important perspectives relative to formula and/or breast feeding with/without high calorie supplements during the first year.

Part I of the Trial is enrollment from birth with collection of blood, urine and umbilical cords for histomorphometry.

Part II will be the "call-back" at 6 to 10 years of age for follow-up assessment of anthropometric and kidney growth, blood pressure and kidney function.

ELIGIBILITY:
Inclusion Criteria:

Stable preterm infants <37 weeks' gestational age; Stable term infants >37 weeks' gestational age

Exclusion Criteria:

<24 weeks gestational age; <600 grams Any anomalies of the genital-urinary or gastrointestinal tract

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants from 24 to 37 weeks' gestation enrolled at birth to be studied for kidney size and function. Term infants >37 weeks' gestation who are stable without complications to serve as controls. Follow-up of preterm and term birth cohort(s) at 6-10 years of age.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-07-23 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in total kidney volume (TKV) from birth to 10 years | Birth, 1 year, 2 years, 6 years, 10 years
  TKV will be measured by 2-D and 3-D renal ultrasound

SECONDARY OUTCOMES:
Development of Hypertension | 1 year, 2 years, 6 years, 10 years
  Blood pressure measurements by sphygmomanometer
Vascular density | 1 year, 2 years, 6 years, 10 years
  Capillary density/ rarefaction to be measured via capillaroscopy
Vascular stiffness | 1 year, 2 years, 6 years, 10 years
  Vascular stiffness measured as pulse wave velocity by tonometry
Change in estimated glomerular filtration rate (eGFR) from birth to 2 years | Birth, 1 year, 2 years, 6 years, 10 years
  Estimated GFR will be calculated from serum creatinine and Cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Marissa J DeFreitas, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami/ Holtz Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abitbol CL, Seeherunvong W, Galarza MG, Katsoufis C, Francoeur D, Defreitas M, Edwards-Richards A, Master Sankar Raj V, Chandar J, Duara S, Yasin S, Zilleruelo G. Neonatal kidney size and function in preterm infants: what is a true estimate of glomerular filtration rate? J Pediatr. 2014 May;164(5):1026-1031.e2. doi: 10.1016/j.jpeds.2014.01.044. Epub 2014 Mar 5. PMID 24607244
- [Result] DeFreitas MJ, Seeherunvong W, Katsoufis CP, RamachandraRao S, Duara S, Yasin S, Zilleruelo G, Rodriguez MM, Abitbol CL. Longitudinal patterns of urine biomarkers in infants across gestational ages. Pediatr Nephrol. 2016 Jul;31(7):1179-88. doi: 10.1007/s00467-016-3327-3. Epub 2016 Feb 9. PMID 26862052
- [Result] DeFreitas MJ, Mathur D, Seeherunvong W, Cano T, Katsoufis CP, Duara S, Yasin S, Zilleruelo G, Rodriguez MM, Abitbol CL. Umbilical artery histomorphometry: a link between the intrauterine environment and kidney development. J Dev Orig Health Dis. 2017 Jun;8(3):349-356. doi: 10.1017/S2040174417000113. Epub 2017 Mar 6. PMID 28260559